CLINICAL TRIAL: NCT04903158
Title: A Single-Center, Single-Dose, Randomized, Open-Label, Parallel Study of Relative Bioavailability With Oral Administration of New and Old Formulations of SHR3680 Tablets in Healthy Male Subjects Under Fasting Conditions
Brief Title: Relative Bioavailability Study of SHR3680
Acronym: SHR-3680
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR3680-BA
Record Dates: First submitted 2021-05-06; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Test formulation of SHR3680
  Interventions: Drug: test SHR3680 tablets
- Reference group (Other): Reference formulation of SHR3680.
  Interventions: Drug: reference SHR3680 tablets

INTERVENTIONS:
Drug: test SHR3680 tablets — Subjects receiving a single oral dose of SHR3680 tablets with 240mg (80mg*3)
  Arms: Test group
Drug: reference SHR3680 tablets — subjects receiving a single oral dose of SHR3680 tablets with 240mg (100mg*2+20mg*2).
  Arms: Reference group

SUMMARY:
This is a single-center, single-dose, randomized, open-label, parallel sstudy to evaluate the relative bioavailability of new and old formulations of SHR3680 tablets in healthy male subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent, and less than 10-year between minimum age and maximum age of the whole subjects;
4. Body weight ≥ 50 kg, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);
5. Agreement to avoid sperm donation for 3 months days after the dose of SHR3680;
6. Glomerular filtration rate (GFR) ≥ 90mL / min / 1.73m2 (see Appendix 1 of the clinical trial protocol for the calculation formula of GFR);

Exclusion Criteria:

1. Any history of epilepsy, including childhood febrile seizures, loss of consciousness, transient ischemic attacks or any conditions that may lead to seizures, such as cerebrovascular disease, brain injury, stroke or brain cancer, etc;
2. Any subject who had any clinically significant acute diseases within one month before screening, including fever or fever as his clinical symptoms, virus, bacteria (including upper respiratory tract infection) or fungi (non-skin) infections;
3. Loss of more than 400 mL blood during the 3 months before the trial (eg, as a blood donor);
4. Allergic constitution;
5. History of drug use, or drug abuse screening positive;
6. Alcoholic or often drinkers;
7. A smoker with 5 cigarettes per day for more than 90 days;
8. Positive serology for hepatitis B surface antigen (HBsAg) and HCV (healthy participants), anti-treponema pallidum virus (TP), or antihuman immunodeficiency virus (HIV) Type 1 and Type 2 (all subjects);
9. Use of any drugs or substances known to be inhibitors or inducers of CYP enzymes within 90 days from the first dose or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to SHR3680 administration and during the study.
10. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
11. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.
12. From 48 hours before taking the study drug to the end of the study, any subject refused to stop using any drinks containing methylxanthine (such as coffee, tea, cola, chocolate, etc.), alcoholic drinks and any fruit juice; they took drinks or foods containing grapefruit 7 days before the first administration of the study drug;
13. Those who received vaccination within 3 months before screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Fr | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
  Fr=AUC (test formulation)/AUC (reference formulation)
Cmax | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
AUC0-t | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
AUC0-∞ | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing

SECONDARY OUTCOMES:
Tmax | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
T1/2 | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
Vd | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
CL/F | predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 and 336 hour after dosing
The incidence and severity of adverse events/serious adverse events (based on NCI-CTCAE 5.0) | From the screening to the scheduled last visit day (Day 49±1 after dosing)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China